CLINICAL TRIAL: NCT02294721
Title: Quality of Pediatric Chest Compression: Comparing Four CPR Feedback Devices With Standard BLS by a Single Rescuer: A Randomised Controlled Manikin Trial
Brief Title: Pediatric Resuscitation With Feedback Devices
Acronym: CPR_NURSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR/2014/10
Record Dates: First submitted 2014-11-16; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without feedback (Experimental): Participants compress the chest of the manikin without CPR feedback device
  Interventions: Device: Standard BLS
- With feedback (Experimental): Participants compress the chest of the manikin with CPR feedback device.
  Interventions: Device: The CPREazy; Device: TrueCPR; Device: The CPR PRO APP; Device: The CardioPump

INTERVENTIONS:
Device: Standard BLS — Resuscitation without feedback devices, standard manual standard basic life support
  Arms: Without feedback
Device: The CPREazy — feedback device-1
  Arms: With feedback
Device: TrueCPR — feedback device -2
  Arms: With feedback
Device: The CPR PRO APP — feedback device -3
  Arms: With feedback
Device: The CardioPump — feedback device- 4
  Arms: With feedback

SUMMARY:
The aim of this study was to compare four different CPR feedback devices to standard BLS in terms of the quality of single rescuer pediatric resuscitation. Therefore, the investigators hypothesis was that there would be no difference between CPR methods in terms of chest compression quality parameters.

DETAILED DESCRIPTION:
Cardiac arrest is a leading cause of death worldwide. High-quality chest compressions are of paramount importance for survival and good neurological outcome. Unfortunately, even health professionals have difficulty performing effective CPR. Chest compression (CC) is often too shallow, compression ratio is inadequate, and hands-off time is too long. CPR feedback devices might be an option for rescuers to in order to increase CC efficiency.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* medical profession (nurses)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Effective compressions | 1 day
  Effective compressions was defined as compression with correct depth (40-50mm), correct hand position and complete decompressions

SECONDARY OUTCOMES:
Chest compression depth | 1 day
  To measure chest compression depth during 8 minutes. Chest compression depth will be measured using the software connected to the manikin and computer
Chest compression rate | 1 day
  To measure the chest compression rate during 8 minutes. Chest compression rate will be measured using the software connected to the manikin and computer
effective compressions ratio | 1day
  effective compressions ratio was defined as effective compressions [%] multiplied by flow time [%]
Flow time was defined as the sum of all periods during which chest compressions were performed | 1 day
  flow time was defined as the sum of all periods during which chest compressions were performed.
absolute hands-off time | 1 day
  absolute hands-off time (HOT) was defined as the sum of all periods without chest compressions or ventilation
VAS (visual analogue scale) | 1 day
  after having completed the 8 min testing period, the study participants were asked how challenging they had experienced standard BLS or resuscitation which the respective feedback device. answers were rated on a 10-point Lickert scale (most difficult = 1 to easiest = 10)
Prefered CPR device | 1 day
  after having completed the 8 min testing period, the study participants were asked how chellenging whitch method they would preferred. answers were rated on a 10-point Lickert scale (lower preferred = 1 to most preferred = 10)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland